CLINICAL TRIAL: NCT06753487
Title: "Effects of Facilitated Postional Release Technique( FPRT) Vs Manual Myofascial Release Technique in Female Patients With Piriformis Syndrome
Brief Title: "Effects of Facilitated Positional Release Technique( FPRT) Vs. Manual Myofascial Release Technique in Female Patients With Piriformis Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/55
Record Dates: First submitted 2024-12-03; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FPRT Group (Experimental): On group A we will perform FACILITATED POSITIONAL RELEASE TECHNIQUE:
  we perform this technique on tight PIRIFORMIS muscle.
  Interventions: Procedure: Facilitated positional release technique
- Myofascial Release technique Group (Active Comparator): On group B we perform MANUAL MYOFASCIAL RELEASE TECHNIQUE on tight PIRIFORMIS muscle same as group A
  Interventions: Procedure: Myofacial Release

INTERVENTIONS:
Procedure: Myofacial Release — Manual Myofascial Release:
  Control group will receive 3- 5 repetitions of Manual Myofascial Release in Piriformis muscle i.e giving ischemic pressure on muscle directly for 90 secs and then release.
  Arms: Myofascial Release technique Group
Procedure: Facilitated positional release technique — FPRT:
  Treatment group will receive 5 repetitions of FACILITATED POSITIONAL RELEASE technique i.e applying pressure over tender area of muscle while maintaining specific postion
  Arms: FPRT Group

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine the "Effects of Facilitated Postional Release Technique( FPRT) Vs Manual Myofascial Release Technique in Female Patients With Piriformis Syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to determine the "Effects of Facilitated positional release technique vs manual myofascial release technique in female patietns with piriformis syndrome.

we make 2 groups control and treatment group . we give FPRT technique to treatment group and manual release technique to control group in patients with piriformis syndrome.

first we take base line readings of HIP ROMS( abduction, adduction, internal rotation, external rotation),NPRS and LEFS(lower extremity functional scale)..

after 2 weeks of treatment again we take same readings and compare both readings.

ELIGIBILITY:
Inclusion Criteria:

* patients with Piriformis syndrome
* 25-50 years
* Only females
* Diagnosed piriformis syndromr
* Pain from 2 months

Exclusion criteria:

* Lumbar Radiculopathy
* Fracture
* trauma to lumbar spine
* surgery/ total hip relpacement
* hip OA

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in ROM | 2 weeks
  Using a Goniometer, specific Hip range of motions (hip abduction, adduction, internal rotation, ext.rotation) will be measured. This process involves positioning the patient in standarized position (i-e supine lying for hip adduction,abduction and sitting for external and internal rotation) aligning the fulcrum of goniometer along the hip axis of motion and recording the readings( in degrees, starts from zero and goes upto the maximum possible acheived range) when joint moves through range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan